CLINICAL TRIAL: NCT07243262
Title: Volatile Organic Compound Assessment in Pancreatic Ductal Adenocarcinoma (VAPOR2)
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Pancreatic Cancer UK (Other); Imperial College Healthcare NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Sherwood Forest Hospitals NHS Foundation Trust (Other); Dorset County Hospital NHS Foundation Trust (Other Government); Buckinghamshire Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 177986
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: Volatile organic compounds (VOCs); Breath analysis; Volatolomics; Validation; Early detection of cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAPOR2 Participants: 6079 participants above the age of 18 years with potential underlying pancreatic cancer referred from primary care according to urgent suspected cancer referral guidelines or referred directly to a pancreatic cancer multidisciplinary team meeting.
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — All participants will fast for a minimum of six hours prior to breath collection. For participants undergoing a procedure, breath samples must be obtained prior to administration of sedation, anaesthetic or other pharmacological agents. After providing written informed consent, participants will be asked to rinse their mouth with water and then provide a breath sample by exhaling into single-use breath collection bags via a mouthpiece that is subsequently sealed.

SUMMARY:
The investigators are developing a non-invasive breath test to help us detect pancreatic cancer earlier. The test detects small molecules called volatile organic compounds that are made by pancreatic cancers.

Pancreatic cancer is a rare disease but patients are often diagnosed at a late stage because their symptoms are the same as those of many common illnesses. This makes it hard for doctors to know which patients need to be tested for pancreatic cancer. If the investigators find pancreatic cancer at a late stage, it reduces the number of treatment choices for patients.

Our test could be offered to patients who are experiencing vague symptoms, which might be caused either by pancreatic cancer or a common illness. This test could help doctors to identify which of those patients may have pancreatic cancer, and ensure they get referred for specialised pancreatic cancer tests. The investigators hope that this will allow us to diagnose pancreatic cancer earlier, increasing treatment choices for patients and improving survival from pancreatic cancer.

The investigators have previously conducted a study (VAPOR1) which collected breath samples from people with and without pancreatic cancer. When the investigators analysed these samples, they found that there is a difference in the volatile organic compounds breathed out by people who have pancreatic cancer compared to those that do not. The investigators used these 'markers' to develop a breath test to diagnose pancreatic cancer. In VAPOR2, the investigators will study our breath test in a much larger group of patients who have been referred for further investigations for potential underlying pancreatic cancer to see how accurately it can pick up the small percentage of people who have pancreatic cancer.

DETAILED DESCRIPTION:
A multicentre double-blind external validation study to validate the breath test to detect PDAC in 6079 adult participants referred from primary care with potential underlying pancreatic cancer, whereby the VOC analyst in the laboratory and the statistician and bioinformatician classifying the VOC profile into cancer/no-cancer will be blinded to the definitive diagnosis of cancer/no-cancer at the time of analysis. Additionally, the radiologist and/or pathologist reporting the reference test (CT, MRI, biopsy) will not have access to the breath test results at any point. Breath test analysis and definitive diagnoses will be held in separate datasets, which will be cleaned and locked before being combined for analysis. The lead statistician will be unblinded at the interim analysis and at the end of the study after the final database lock once all the study data has been collected and cleaned, to calculate the accuracy of the prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥ 18 years old
* Referral from primary care according to the urgent suspected cancer referral guidelines for potential underlying pancreatic cancer, or referral directly to a pancreatic cancer multidisciplinary team meeting

Exclusion Criteria:

* Previous pancreatic resection
* History of another cancer (other than non-melanoma skin cancers) within three years
* Pregnant participants (pregnancy status to be confirmed verbally with the participant)
* Participants with co-morbidities preventing breath collection
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants above the age of 18 years with potential underlying pancreatic cancer referred from primary care according to urgent suspected cancer referral guidelines will be invited to participate in the study. In addition, participants referred directly to a pancreatic cancer multidisciplinary team meeting will also be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 6079 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Validation of a triage breath test for detecting pancreatic ductal adenocarcinoma in 6079 participants referred from primary care with potential underlying pancreatic cancer. | 36 months
  Estimation of sensitivity, specificity and numbers of false positives (with 95% confidence intervals) for a breath test to detect pancreatic ductal adenocarcinoma

SECONDARY OUTCOMES:
To test feasibility of the breath test in a large population | 36 months
  Feasibility of the breath test in a large population will be reported as the proportion of tests that were completed and analysed.
Economic modelling for scaling up breath testing into clinical practice. | 36 months
  To assess the cost-benefit trade-offs of using the breath test in the symptomatic population referred for suspicion of PDAC. To inform its utilisation within the NHS, the specific objectives are to:
  (i) map out current and breath test-assisted clinical pathways for PDAC referrals; (ii) estimate the health economic impact for the NHS by adopting the augmented breath test; and (iii) consider barriers to adoption and develop mitigation strategies for scaling-up in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Professor George B Hanna, PhD, FRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No